CLINICAL TRIAL: NCT06818357
Title: Sensory Perception in Children With Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-8
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy; Sensory Disorders; Perception Disorders
Keywords: epilepsy; Sensory Disorders; Perception Disorders
MeSH Terms: conditions — Epilepsy; Sensation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children diagnosed with epilepsy
- Control group: healthy children

SUMMARY:
Epilepsy is a chronic neurological disorder characterized by abnormal neuronal activity, affecting approximately 0.5-1% of children worldwide. It has significant social, psychological, and physical consequences, leading to impairments in cognitive, motor, and behavioral functions. Sensory processing disorders (SPDs) further contribute to these challenges, affecting children's ability to regulate and interpret sensory information, which impacts learning, daily functioning, and emotional regulation.

SPDs are categorized into sensory modulation disorder, sensory-based motor disorder, and sensory discrimination disorder. Dunn's sensory processing model identifies four sensory profiles: low registration, sensory seeking, sensory sensitivity, and sensory avoidance. Sensory modulation disorders, including sensory over-responsivity, under-responsivity, and seeking behaviors, can contribute to behavioral and functional difficulties in children with epilepsy.

Existing studies on sensory processing in children with epilepsy are limited by small sample sizes and non-comprehensive assessments. This study aims to investigate sensory profiles and perception in a larger sample to enhance early detection and intervention strategies.

Objectives:

Evaluate sensory perception in children with epilepsy. Examine sensory profiles within this population. The study will include children aged 2-17 years meeting specific criteria. Data collection will involve demographic and epilepsy-related information (seizure onset, frequency, medication, comorbidities). A neurology specialist will assess cerebellar pathology. Sensory processing will be evaluated using the Sensory Processing Measure (SPM), a validated tool assessing sensory processing, balance, body awareness, ideation, and social participation.

Based on prior studies, the required sample size is 34 participants. Statistical analyses will be performed using IBM SPSS v.26.0 and R v4.3.0. Normality will be assessed through graphical and statistical tests. Independent samples t-tests, Mann-Whitney U tests, chi-square tests, and correlation analyses will be applied where appropriate. The significance level is set at p<0.05.

This study will contribute to the understanding of sensory perception in children with epilepsy, addressing gaps in the literature and supporting clinical interventions to improve their daily functioning and well-being.

DETAILED DESCRIPTION:
Epilepsy is a transient condition that occurs due to abnormal high neuronal activity or asynchronous neuronal circuits in the brain and is defined as such by the International League Against Epilepsy (ILAE). Epilepsy is one of the most common chronic childhood diseases, affecting approximately 0.5-1% of children worldwide. According to the relevant literature, an estimated 10.5 million children under the age of 15 are currently diagnosed with active epilepsy. Epilepsy is classified based on clinical characteristics such as seizure type, age of onset, cognitive and developmental history, presence of neurological symptoms, family history, electroencephalography findings, seizure triggers, seizure occurrence during sleep, and prognosis.

Seizures in children with epilepsy have profound negative effects on social, psychological, and physical health, leading to impairments in cognitive functioning. Various studies have reported potential deficits in intelligence, memory, learning, attention, motor skills, and behavioral abilities in children with epilepsy. Additionally, deficits in executive functions and motor coordination, along with difficulties in responding to environmental demands, have been reported.

Beyond epilepsy, sensory processing disorders significantly impact children's ability to process, regulate, and interpret sensory information from the environment. These disorders affect cognitive, motor, behavioral, and emotional responses. Sensory processing disorders are commonly associated with impairments in neuropsychomotor development. Children experiencing these difficulties may exhibit behavioral issues, sleep disorders, social interaction challenges, and aggression. Additionally, heightened emotional reactions and frequent crying are commonly observed behavioral traits. Sensory processing disorders can negatively affect self-regulation, learning, functional behaviors, daily living skills, motor organization, and school performance.

Sensory processing disorders are typically classified into three main categories: sensory modulation disorder, sensory-based motor disorder, and sensory discrimination disorder. According to Dunn's sensory processing theory, individuals' responses to sensory stimuli vary based on their neurological threshold levels and their type of response to stimuli. Dunn describes a continuous interaction in which individuals' responses to sensory stimuli may lead to maladaptive behaviors. Dunn classifies these responses into passive and active self-regulation strategies. Passive self-regulation allows individuals to experience sensory stimuli without controlling them, whereas active self-regulation involves controlling and modulating stimuli. Based on these mechanisms, four distinct sensory profiles are defined: low registration, sensory seeking, sensory sensitivity, and sensory avoidance.

Low registration refers to a high neurological threshold, resulting in individuals not noticing sensory stimuli or responding very slowly. Sensory seeking describes individuals with a high neurological threshold who actively seek excessive sensory input. In this case, individuals may be drawn to strong stimuli such as intense smells, sounds, or lights. Sensory sensitivity is characterized by a low sensory threshold, where individuals exhibit heightened sensitivity to environmental stimuli but do not generate an active response. Sensory avoidance, also associated with a low sensory threshold, involves active strategies to avoid distressing stimuli.

Sensory modulation disorders involve difficulties in detecting, regulating, and interpreting sensory stimuli or in generating appropriate responses to them. In the literature, sensory modulation disorders are classified into three main categories: sensory over-responsivity, sensory under-responsivity, and sensory seeking. These disorders may lead to behavioral problems due to an inability to regulate responses to environmental sensory stimuli.

Studies conducted on children with epilepsy have generally focused on small sample sizes and specific epilepsy types, using short-form sensory profile assessments. Moreover, most of these studies have included a limited number of participants. Despite these limitations, existing research highlights the need for further investigation into the prevalence and effects of sensory modulation and perception disorders in children with epilepsy.

The aim of this study is to investigate the sensory profiles of children with epilepsy in a larger sample and identify the presence of sensory perception disorders in this population. By doing so, this study aims to improve the understanding of sensory processing disorders in children with epilepsy and contribute to the development of effective early detection methods. This research will facilitate a more detailed identification of sensory perception disorders among children with epilepsy, addressing gaps in the literature and supporting necessary interventions to enhance their daily living skills and overall health.

Objectives:

To evaluate sensory perception in children with epilepsy.

To examine the sensory profiles of children with epilepsy.

If significant results are obtained, these findings are intended to contribute to clinical practice and scientific research. The study will be conducted with children aged 2-17 years who meet the inclusion criteria and whose families voluntarily agree to participate. During the study period, eligible children will be assessed according to inclusion criteria. Detailed demographic information and epilepsy-related characteristics will be collected, including the age of seizure onset, seizure frequency, medications used, comorbid conditions, and family psychiatric history. A neurology specialist will assess the presence of cerebellar pathology in the participating children. Sensory perception will be evaluated using the Sensory Processing Measure.

Sensory Processing Measure

The Sensory Processing Measure (SPM) is designed to assess children aged 5-12 years. It is a standardized caregiver-report tool that evaluates behaviors related to sensory processing, balance, body awareness, ideation, and social participation. Compared to sensory profiles, the SPM assesses different aspects of sensory processing (e.g., perception and discrimination) and their impact on social participation. It is an effective tool for distinguishing sensory processing characteristics between children with different diagnoses and typically developing children. The scale consists of 75 items and includes eight subdomains:

Social participation (items 1-10)

Vision (items 11-21)

Hearing (items 22-29)

Touch (items 30-40)

Taste/smell (items 41-45)

Body awareness (items 46-55)

Balance and movement (items 56-66)

Planning and ideas (items 67-75)

The scale is Likert-type, with response options as follows: 1 (never), 2 (sometimes), 3 (frequently), and 4 (always). The Turkish validity and reliability study of the scale was conducted by Özbakır.

A literature review revealed that no direct studies have examined sensory perception in this specific population. However, previous studies have suggested that sensory perception and sensory modulation may yield similar results. Based on this, a study measuring sensory perception was considered. In that study, a large effect size (d=1.31) was observed between patient and control groups. Using this effect size, the required sample size was calculated for an independent samples t-test with 90% power and a 5% error rate. The analysis determined that at least 14 participants per group (a total of 28) were necessary. Assuming a 20% attrition rate, the final target sample size was set at a minimum of 34 participants (17 per group). The calculation was performed using G-Power 3.1.9.7 software.

Statistical analyses will be conducted using IBM SPSS Statistics v.26.0 (Armonk, NY: IBM) and R Statistical Software (v4.3.0; R Core Team 2023). Descriptive statistics will be reported as means and standard deviations for numerical data, or quartiles where applicable, and as counts and percentages for categorical data. Normality assumptions will be checked using graphical methods (QQ plots, histograms) and hypothesis tests (Shapiro-Wilk test). Independent samples t-tests will be used for comparing numerical variables between groups when assumptions are met; otherwise, the Mann-Whitney U test will be applied. Categorical variable comparisons will be conducted using chi-square tests (Pearson, Yates, Fisher's Exact Test). Correlations between numerical variables will be analyzed using Pearson or Spearman correlation coefficients depending on assumption fulfillment. The significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of epilepsy Having had an epileptic seizure within the year before the data collection period Being between the ages of 2 and 17 Voluntarily agreeing to participate in the study

Exclusion Criteria:

cerebral palsy, hydrocephalus, autism spectrum disorder, pervasive developmental disorder, learning disability, dyslexia, genetic disease, metabolic disease, neuromuscular disease.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children diagnosed with epilepsy and healthy children
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensory Processing Measure | 1 year
  Sensory Processing Measure
  The Sensory Processing Measure (SPM) is designed to assess children aged 5-12 years. It is a standardized caregiver-report tool that evaluates behaviors related to sensory processing, balance, body awareness, ideation, and social participation. Compared to sensory profiles, the SPM assesses different aspects of sensory processing (e.g., perception and discrimination) and their impact on social participation. It is an effective tool for distinguishing sensory processing characteristics between children with different diagnoses and typically developing children. The scale consists of 75 items and includes eight subdomains:
  Social participation (items 1-10)
  Vision (items 11-21)
  Hearing (items 22-29)
  Touch (items 30-40)
  Taste/smell (items 41-45)
  Body awareness (items 46-55)
  Balance and movement (items 56-66)
  Planning and ideas (items 67-75)
  The scale is Likert-type, with response options as follows: 1 (never), 2 (sometimes), 3 (frequently), and 4 (alwa

CONTACTS AND LOCATIONS:
Overall Officials: Seda AYAZ TAS, PhD, Study Director — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] van Campen JS, Jansen FE, Kleinrensink NJ, Joels M, Braun KP, Bruining H. Sensory modulation disorders in childhood epilepsy. J Neurodev Disord. 2015;7:34. doi: 10.1186/s11689-015-9130-9. Epub 2015 Oct 23. PMID 26504494